CLINICAL TRIAL: NCT04435860
Title: Evaluation of Relationship Between Trunk, Proximal Girdle Muscles' Strength, and Functionality and Disease Activity in Male Patients With Ankylosing Spondylitis
Brief Title: Muscle Strength Evaluations in Ankylosing Spondylitis
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-08/115
Record Dates: First submitted 2020-06-15; First posted 2020-06-17 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Ankylosing Spondylitis
Keywords: Muscle Powers; Functionality; Disease Activity
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ankylosing Spondylitis: Patients with ankylosing spondylitis meeting the inclusion and exclusion criteria
  Interventions: Other: Truncal flexion-extension muscle power; Other: Truncal extension muscle power; Other: Cervical flexion muscle power; Other: Cervical extension muscle power; Other: Cervical lateral flexion muscle powers; Other: Shoulder flexion muscle power; Other: Shoulder extension muscle power; Other: Shoulder internal rotation muscle power; Other: Shoulder external rotation muscle power; Other: Shoulder abduction muscle power; Other: Hip flexion muscle power; Other: Hip extension muscle power; Other: Hip abduction muscle power; Other: Hip internal rotation muscle power; Other: Hip external rotation muscle power; Other: Bath Ankylosing Spondylitis Functional Index (BASFI); Other: Bath Ankylosing Spondylitis Disease Activity Index (BASDAI); Other: The Health assessment questionnaire (HAQ); Other: Bath Ankylosing Spondylitis Metrology Index (BASMI)
- Healthy Controls: Healthy individuals meeting the exclusion criteria
  Interventions: Other: Truncal flexion-extension muscle power; Other: Truncal extension muscle power; Other: Cervical flexion muscle power; Other: Cervical extension muscle power; Other: Cervical lateral flexion muscle powers; Other: Shoulder flexion muscle power; Other: Shoulder extension muscle power; Other: Shoulder internal rotation muscle power; Other: Shoulder external rotation muscle power; Other: Shoulder abduction muscle power; Other: Hip flexion muscle power; Other: Hip extension muscle power; Other: Hip abduction muscle power; Other: Hip internal rotation muscle power; Other: Hip external rotation muscle power

INTERVENTIONS:
Other: Truncal flexion-extension muscle power — Patient performs a maximum truncal flexion laying supine on the bed with cap of muscle tester placed on sternum,
Other: Truncal extension muscle power — Patient performs a maximum truncal extension laying prone on the bed while the cap of manual muscle tester placed on vertebrae at the level of midline between superior angles of scapulae.
Other: Cervical flexion muscle power — Patient performs a maximum cervical flexion sitting while the cap of manual muscle tester placed on the middle of the forehead.
Other: Cervical extension muscle power — Patient performs a maximum cervical extension sitting while the cap of manual muscle tester placed on protuberantia occipitalis.
Other: Cervical lateral flexion muscle powers — Patient performs a maximum cervical lateral flexions on right and left sitting while the cap of manual muscle tester placed on relevant pterion.
Other: Shoulder flexion muscle power — Patient performs a maximum shoulder flexion of the dominant side on upright while the cap of manual muscle tester placed on midpoint of the line between anterior aspect of acromion and anterior elbow.
Other: Shoulder extension muscle power — Patient performs a maximum shoulder flexion of the dominant side on upright while the cap of manual muscle tester placed on midpoint of the line between posterior aspect of acromion and posterior elbow.
Other: Shoulder internal rotation muscle power — Patient performs a maximum shoulder internal rotation of the dominant side on upright while the cap of manual muscle tester placed on midpoint of the line between anterior elbow and wrist.
Other: Shoulder external rotation muscle power — Patient performs a maximum shoulder external rotation of the dominant side on upright while the cap of manual muscle tester placed on midpoint of the line between posterior elbow and wrist.
Other: Shoulder abduction muscle power — Patient performs a maximum shoulder abduction of the dominant side on upright while the cap of manual muscle tester placed on midpoint of the line lateral aspect of acromion and lateral epicondyle.
Other: Hip flexion muscle power — Patient performs a maximum hip flexion laying supine on the bed while the cap of manual muscle tester placed on middle of the anterior thigh.
Other: Hip extension muscle power — Patient performs a maximum hip extension laying prone on the bed while the cap of manual muscle tester placed on middle of the posterior thigh.
Other: Hip abduction muscle power — Patient performs a maximum hip abduction laying supine on the bed while the cap of manual muscle tester placed on middle of the lateral thigh.
Other: Hip internal rotation muscle power — Patient performs a maximum hip internal rotation laying supine on the bed while the cap of manual muscle tester placed on the midline between lateral condyle of femur and lateral malleolus.
Other: Hip external rotation muscle power — Patient performs a maximum hip external rotation laying supine on the bed while the cap of manual muscle tester placed on the midline between medial condyle of femur and medial malleolus.
Other: Bath Ankylosing Spondylitis Functional Index (BASFI) — This questionnaire evaluates the functionality in patients with AS. The ten questions that comprise the BASFI were chosen with input from patients with AS. The first 8 questions evaluate activities related to functional anatomical limitations due to the course of this inflammatory disease. The final 2 questions evaluate the patients' ability to cope with everyday life. A visual analogue scale (with 0 being "easy" and 10 "impossible) is used to answer the questions on the test. The final score varies between 0 and 10.
  Groups: Ankylosing Spondylitis
Other: Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) — This questionnaire evaluates the disease activity level in patients with AS. The BASDAI consists of a 0 - 10 scale measuring discomfort, pain, and fatigue (0 being no problem and 10 being the worst problem) in response to six questions asked of the patient pertaining to the five major symptoms of AS. The final score varies between 0 and 10.
  Groups: Ankylosing Spondylitis
Other: The Health assessment questionnaire (HAQ) — The Health assessment questionnaire (HAQ) is a questionnaire for the assessment of disability in an individual. The patients report the amount of difficulty they have in performing eight daily living activities. Each question asks on a scale ranging from 0 to 3 if the categories can be performed without any difficulty (scale 0) up to cannot be done at all (scale 3). The final score varies between 0 and 3.
  Groups: Ankylosing Spondylitis
Other: Bath Ankylosing Spondylitis Metrology Index (BASMI) — Bath Ankylosing Spondylitis Metrology Index, a combined index to assess the spinal mobility. It evaluates the patients regarding cervical rotation, tragus-to-wall distance, lumbar flexion, lumbar lateral flexion and intermalleolar distance. The total score varies between 5 to 15 in patients with ankylosing spondylitis
  Groups: Ankylosing Spondylitis

SUMMARY:
This study evaluates how the trunk and proximal girdle muscles are affected in male patients with ankylosing spondylitis, compared to healthy controls.

DETAILED DESCRIPTION:
Ankylosing spondylitis is a chronic, inflammatory rheumatic disease with an unclear etiology which causes back pain and affects the functionality of axial skeleton. Besides the effect upon axial skeleton, the disease also affects the peripheral joints. In most patients, tenuous affection of peripheral joints occurs however, in some others the disease causes impaired spinal mobility and articular instability. This causes proximal girdle muscles and trunk muscles of the patients to be exposed to excessively stress and in conclusion deformities develop. Maximum force generated by a muscle or muscle group directly effects the physical ability of an individual, and manual muscle dynamometers are used to directly evaluate the muscle strength. In this manner the investigators aim to evaluate trunk and proximal girdle muscles' powers in male patients with ankylosing spondylitis and analyze the correlation between muscle powers, and functionality and disease activity.

ELIGIBILITY:
Inclusion Criteria:

1. Having a diagnosis of ankylosing spondylitis according to Modified NewYork criteria
2. Being male
3. Aged ≥18

Exclusion Criteria:

1. Severe cardiac or pulmonary or renal disease
2. Accompanying fibromyalgia
3. Severe psychiatric disorder
4. Other disease limiting spinal, shoulder or hip range of motion
5. Myopathy, neuropathy or radiculopathy that may cause muscle weakness
6. Using high dose steroids
7. Endocrinological disorders
8. Malignancy
9. Pregnancy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Controls: Healthy volunteers meeting inclusion criteria accepting to participate Ankylosing spondylitis group: Ankylosing spondylitis patients meeting inclusion criteria accepting to participate
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2020-09-04 (Actual); Study Completion 2020-09-04 (Actual)

PRIMARY OUTCOMES:
Cervical muscle powers | 1 day
  Cervical flexion, extension, and lateral flexion muscle powers in kilograms as assessed with handheld dynamometer.
Truncal muscle powers | 1 day
  Truncal flexion and extension muscle powers in kilograms as assessed with handheld dynamometer.
Shoulder girdle muscle powers | 1 day
  Shoulder flexion, extension, abduction, internal rotation, and external rotation muscle powers in kilograms as assessed with handheld dynamometer.
Hip girdle muscle powers | 1 day
  Hip flexion, extension, abduction, internal rotation, and external rotation muscle powers in kilograms as assessed with handheld dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: Ozan Volkan Yurdakul, Assoc Prof, Principal Investigator — Bezmialem University
Locations (1):
- Bezmialem University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim SC, Lee YG, Park SB, Kim TH, Lee KH. Muscle Mass, Strength, Mobility, Quality of Life, and Disease Severity in Ankylosing Spondylitis Patients: A Preliminary Study. Ann Rehabil Med. 2017 Dec;41(6):990-997. doi: 10.5535/arm.2017.41.6.990. Epub 2017 Dec 28. PMID 29354575
- [Background] Daloia LMT, Leonardi-Figueiredo MM, Martinez EZ, Mattiello-Sverzut AC. Isometric muscle strength in children and adolescents using Handheld dynamometry: reliability and normative data for the Brazilian population. Braz J Phys Ther. 2018 Nov-Dec;22(6):474-483. doi: 10.1016/j.bjpt.2018.04.006. Epub 2018 May 4. PMID 29802034
- [Background] De Blaiser C, De Ridder R, Willems T, Danneels L, Roosen P. Reliability and validity of trunk flexor and trunk extensor strength measurements using handheld dynamometry in a healthy athletic population. Phys Ther Sport. 2018 Nov;34:180-186. doi: 10.1016/j.ptsp.2018.10.005. Epub 2018 Oct 12. PMID 30366246
- [Derived] Yurdakul OV, Ince OE, Bagcier F, Kara M, Kultur E, Aydin T. Evaluating the strength of spinal and proximal girdle muscles in patients with axial spondyloarthritis: Correlation with activity, disability, and functionality. Int J Rheum Dis. 2021 May;24(5):701-710. doi: 10.1111/1756-185X.14102. Epub 2021 Mar 22. PMID 33750032